CLINICAL TRIAL: NCT03073629
Title: Implementation of a Clinical Pathway to Improve Outcomes in Emergency Department Patients With Right Ventricular Failure
Brief Title: Assessing Outcomes in ED Patients With RV Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Found not to be feasible
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Frances Russell, Assistant Professor of Emergency Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1605974831
Record Dates: First submitted 2017-03-02; First posted 2017-03-08 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2017-03

CONDITIONS: Right Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Pathway Cohort (Active Comparator): Patients with isolated RV failure will be evaluated and managed in a specialized cardiovascular clinic.
  Interventions: Diagnostic Test: Clinical Pathway
- Standard Care (No Intervention): Patients with isolated RV failure will receive standard care and follow up.

INTERVENTIONS:
Diagnostic Test: Clinical Pathway — Patients will be evaluated and managed in a specialized cardiovascular clinic to determine the etiology of right heart failure and begin treatment.
  Arms: Clinical Pathway Cohort

SUMMARY:
Millions of Americans seek emergency care for acute shortness of breath, and many undergo computerized tomographic pulmonary angiography (CTPA) testing that is negative for acute disease. Management of patients with persistent shortness of breath despite normal testing continues to pose a challenge for clinicians. Right ventricular (RV) failure is a common cause of dyspnea that brings patients to the emergency department (ED), however, it is often not considered in the differential diagnosis, remains unrecognized, or patients are not properly followed up once diagnosed. Delays in diagnosis and management of RV failure are associated with poor outcomes. The investigators propose a novel clinical pathway, which entails identifying and enrolling patients with RV failure in the ED, then referring them to a specialized cardiovascular clinic where they will receive a standardized evaluation and management plan. Our hypothesis is that management of RV failure, through this pathway, will improve patient outcomes when compared to standard care. The primary outcome will assess 1-year unscheduled healthcare visits.

ELIGIBILITY:
Inclusion Criteria:

* adult patients > 18 years old,
* with a non-significant CTPA scan (i.e. no acute disease), dyspnea PLUS an emergency physician performed echocardiogram with isolated RV failure OR CTPA scan with evidence of pulmonary hypertension OR comprehensive echocardiogram within 3 months of index hospital visit showing isolated RV dysfunction

Exclusion Criteria:

* Currently being evaluated and/or treated for RV failure or PH,
* those unable to have a comprehensive echocardiography performed,
* those with indeterminate RV function OR LV dysfunction on comprehensive echocardiography, and
* those patients with circumstances where they may be lost to follow-up (homeless, prisoner, severe psychiatric disorder, no reliable contact information).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
Unscheduled healthcare visits | 1 year

SECONDARY OUTCOMES:
Mortality | 1 year
Hospital re-admissions | 1 year
Change in quality of life via the SF-36 | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Methodist Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No